CLINICAL TRIAL: NCT00994058
Title: Pilot Study to Evaluate A Prototype Electronic Uterine Inhibitor to Prevent Preterm Contractions
Brief Title: Pilot Study of Electronic Uterine Contraction Inhibitor
Acronym: PSEUCI
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The Investigator has changed institutions.
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Graham Gaylord Ashmead, MD, Dept OB/GYN, Winthrop University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 09034
Record Dates: First submitted 2009-10-07; First posted 2009-10-14 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Prematurity
Keywords: Preterm Labor; Uterine Inhibitor; Electro-Inhibition
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intevention with Inhibitor (Experimental)
  Interventions: Device: Electrical Inhibition (EI) Uterine Pacemaker

INTERVENTIONS:
Device: Electrical Inhibition (EI) Uterine Pacemaker — An external powered pulse generator, pacemaker for external stimulation of the uterine muscle through the vaginal canal for the therapeutic use of preventing preterm birth.
  Patients with preterm contractions (< 37 weeks gestation) will be monitored for contraction frequency for 20 minutes before, 20 minutes during use of EI and 20 minutes after EI/uterine inhibitor/pacemaker. Device generates a weak electrical current (0-10mA, 0-50 Hz, 0-50mS).

SUMMARY:
The objective is to test a novel paradigm for the inhibition of human preterm uterine contractions.

The study hypothesis is that human preterm contractions can be safely inhibited with a weak electrical current provided by an electrical inhibition/uterine pacemaker device.

Preterm birth is still a major problem. Current methods of preventing the uterine contractions of preterm are limited and associated with many side-effects affecting both the mother and baby. A reliable method of preventing preterm uterine contractions would be an important discovery. Such a method could eventually lead to a long-term goal of decreasing neonatal morbidity and mortality.

DETAILED DESCRIPTION:
The study design is a Pilot Study to confirm the safety of the uterine inhibitor/pacemaker and measure its effect on women experiencing preterm labor.

A total of 10 (ten) patients will be enrolled in this pilot study to confirm the methodology and safety of the device. Patients who meet the inclusion criteria and none of the exclusion criteria will be recruited for the study.

The study device (EI/uterine inhibitor/pacemaker) has been classified by FDA as an Investigational Device Exemption (IDE) number G080036, Class A device. The EI/uterine inhibitor/pacemaker device is FDA cleared for research of the prevention of the prevention of the human contractions of preterm birth.

This proposal is for an initial prospective FDA approved pilot study. After FDA evaluation of the pilot study findings and approval, the pilot study may lead eventually to a prospective randomized controlled clinical study.

Only adult women who are experiencing uterine contractions due to the birthing process are eligible.

Study patients will be informed about the purpose of the EI/uterine inhibitor/pacemaker device and give informed consent prior to its use. The device will be used for only 20 minutes, preceded and followed by a 20 minute control period.

During the birthing process recordings of the uterine contractions will be recorded. Comparison will be made of these uterine contraction records pre and post use use of the EI/uterine inhibitor/pacemaker device. The uterine contraction tracings will be compared and analyzed for differences in the frequency of contractions.

The patients will also be told how to express the strength of any of their subjective pain in a manner that can be documented in a questionnaire. Study patients will also have their record of the type and amount of pain medication they have received noted on their patient log forms.

RISK:

Previous human and animal studies indicate minimal risk to either baby or mother. Human studies showed no effect on the fetal or maternal heart rate. Real-time monitoring of the fetal and maternal heart rate during the study will protect against there potential risks.

BENEFIT:

Reducing the frequency of preterm uterine contractions is a first step to preventing preterm birth,but the proposed investigation is not, itself, expected to prevent any preterm births. However, the investigation could have great benefit to future mothers and their babies.

ELIGIBILITY:
Inclusion Criteria:

1. 24 to 34 weeks pregnant
2. preterm labor

   * at least one contraction every 5 minutes for 30 minutes
   * > 3 cm cervical dilation; > 80% cervical effacement
3. Have received tocolysis therapy
4. Anticipate a normal spontaneous vaginal delivery (NSVD)
5. Be at least 18 years of age
6. Have signed a written informed consent document
7. Be willing and able to comply with study requirements

Exclusion Criteria:

1. Severe preeclampsia
2. Severe abruption placenta
3. Rupture of amnionic membranes
4. Frank chorioamnionitis
5. Fetal death
6. Fetal anomaly incompatible with life
7. Severe fetal growth restriction (estimated fetal weight <5%)
8. Mature fetal lung studies
9. Maternal cardiac arrythmias
10. A permanent cardiac pacemaker
11. A fetal cardiac arrhythmia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Contraction frequency | 60 minutes

SECONDARY OUTCOMES:
Preterm birth | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Graham G Ashmead, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

REFERENCES:
- [Background] Karsdon J, Garfield RE, Shi SQ, Maner W, Saade G. Electrical inhibition of preterm birth: inhibition of uterine contractility in the rabbit and pup births in the rat. Am J Obstet Gynecol. 2005 Dec;193(6):1986-93. doi: 10.1016/j.ajog.2005.05.009. PMID 16325601